CLINICAL TRIAL: NCT03579966
Title: Long Term Safety Study of Amifampridine Phosphate in Patients With MuSK Antibody Positive and AChR (Acetylcholine Receptor) Antibody Positive Myasthenia Gravis
Brief Title: Long Term Safety Study of Amifampridine Phosphate in MuSK-MG (Muscle Specific Tyrosine Kinase Myasthenia Gravis)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Lack of measure appropriate data (MG-ADL).
Sponsor: Catalyst Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MSK-003
Record Dates: First submitted 2018-06-05; First posted 2018-07-09 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Myasthenia Gravis, MuSK; AChR Myasthenia Gravis
Keywords: Amifampridine Phosphate Amifampridine; 3,4-Diaminopyridine Phosphate; 3,4-Diaminopyridine; 3,4-DAP; Firdapse®; Myasthenia Gravis; MuSK; AChR
MeSH Terms: conditions — Myasthenia Gravis | interventions — Amifampridine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- amifampridine phosphate (Experimental): tablets equivalent to 10mg amifampridine, 3 to 4 times per day. Initially, the daily amifampridine doses were to be the doses that were determined at the end of the Run-in Period from the MSK-002 study. The usual range was from 30 to 80 mg total daily dose, given in three (3) or four (4) doses, with no single dose > 20 mg
  Interventions: Drug: Amifampridine Phosphate

INTERVENTIONS:
Drug: Amifampridine Phosphate — tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day

SUMMARY:
Evaluate the long-term safety of amifampridine phosphate in patients with MuSK antibody positive and AChR antibody positive myasthenia gravis.

DETAILED DESCRIPTION:
The Primary objective :

To characterize the long-term safety and tolerability of amifampridine phosphate in patients with MG

The Secondary Objective:

To assess the clinical efficacy of amifampridine phosphate over time in patients with MG based on change in Myasthenia Gravis Activities of Daily Living Score (MG-ADL)

This was a long-term extension study for subjects who participated in Protocol MSK-002 where the efficacy and safety of amifampridine was evaluated in subjects diagnosed with MuSK MG or AChR-MG. The optimal dose and schedule for amifampridine from the end of the Run-in Period from Study MSK-002 was initially used for each patient. The Investigator could adjust the dose of amifampridine during the course of the trial, in order to optimize neuromuscular benefit for the patient. Clinic visits for safety assessment and for evaluation of MG-ADL were made at Months 3, 6, 9, 12, 15, 21, 27, 33 and 39. Additional visits could occur at the discretion of the Investigator.

The Original protocol (12 Nov 2017) included analysis of MG-ADL change over time, however, Statistical Analysis Plan (SAP), dated 21 Feb 2023, removed the analysis of MG-ADL score change over time.

ELIGIBILITY:
Inclusion Criteria

1. Participated in the MSK-002 study
2. Willing and able to provide written informed consent after the nature of the study has been explained and before the start of any research-related procedures.
3. Female patients of childbearing potential must have a negative pregnancy test (urine human chorionic gonadotropin [HCG] at the end of MSK-002 study); and must practice an effective, reliable contraceptive regimen during the study and for up to 30 days following discontinuation of treatment.
4. Ability to participate in the study based on overall health of the patient and disease prognosis, as applicable, in the opinion of the Investigator; and able to comply with all requirements of the protocol, including completion of study questionnaires.

Individuals who met any of the exclusion criteria in the original protocol or those listed below are not eligible to participate in the study:

1. Epilepsy and currently on medication.
2. Clinically significant abnormalities in 12 lead ECG, in the opinion of the Investigator.
3. Breastfeeding or pregnant at Screening or planning to become pregnant at any time during the study.
4. Intolerable amifampridine-related side effects
5. Treatment with an investigational drug (other than amifampridine) or device while participating in this study.
6. Any medical condition that, in the opinion of the Investigator, might interfere with the patient's participation in the study, poses an added risk for the patient, or confound the assessment of the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2018-06-11 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renato Mantegazza, MD, Principal Investigator — Carlo Besta Neurological Institute
Locations (3):
- United States (2):
  - Cleveland Clinic, Cleveland, Ohio
  - Univerity of Pennsylvania, Philadelphia, Pennsylvania
- Department of Neuroimmunology and Neuromuscular Diseases Carlo Besta Neurological Institute Via Celoria, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: extension study to MSK-002
Period: Overall Study
Arm/Group | Amifampridine Phosphate
Started | 63
Completed | 3
Not Completed | 60
Not completed — Adverse Event | 6
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 10
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 16
Not completed — Study terminated by Sponsor | 22
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Arm/Group | Amifampridine Phosphate
Number analyzed (Participants) | 63
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (14.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 59
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 36
  Italy | 27
Weight [Mean (Standard Deviation); unit: Kg] — Population: Baseline weight not recorded for 4 participants.
  Kg
    number analyzed (Participants) | 59
    (all) | 85.9 (24.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (Safety and Tolerability)
Description: Evaluate the long-term safety and tolerability of amifampridine phosphate through the number of patients with treatment-emergent adverse events mapped to the Medical Dictionary for Regulatory Activities (MedDRA) SOCs and PTs. [ Time Frame: over 39 months ] Descriptive statistics will be used to summarize study data.
Time Frame: over 39 months
Measure: Count of Participants; unit: Participants
Groups:
- Treatment Emergent Adverse Events: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day.
Arm/Group | Treatment Emergent Adverse Events
Number analyzed (Participants) | 63
Participants | 58

ADVERSE EVENTS:
Time Frame: Study Duration 39 months
Description: Serious classification based on the FDA regulatory definition of a serious AE.
Groups:
- Serious Adverse Event: Amifampridine Phosphate: tablets equivalent to 10mg amifampridine, titrated to an efficacious and tolerable dose, 3 to 4 times a day.
Arm/Group | Serious Adverse Event
All-Cause Mortality (participants affected / at risk) | 0/63
Serious Adverse Events (participants affected / at risk) | 14/63
Other Adverse Events (participants affected / at risk) | 58/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serious Adverse Event (N=63)
Aortic Valve Stenosis (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (1)
corona virus infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3)
Staphylococcal infection (Infections and infestations) | 1 (1)
cervical spine stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Myasthenia Gravis (Nervous system disorders) | 4 (4)
Myasthenia Gravis Crisis (Nervous system disorders) | 1 (1)
abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Serious Adverse Event (N=63)
Cataract (Ear and labyrinth disorders) | 4 (4)
Diplopia (Ear and labyrinth disorders) | 3 (3)
Vitreous Floaters (Eye disorders) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Hypoasthesia Oral (Gastrointestinal disorders) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4)
Paresthesia Oral (Gastrointestinal disorders) | 15 (15)
Vomiting (Gastrointestinal disorders) | 4 (4) — Does not include SAE
Asthenia (General disorders) | 4 (4)
Fatigue (General disorders) | 6 (6)
Pyrexia (General disorders) | 3 (3)
Bronchitis (Infections and infestations) | 2 (2)
Corona Virus Infection (Infections and infestations) | 4 (4) — Does not include the SAEs
Nasopharyngitis (Infections and infestations) | 4 (4)
Onychomycosis (Infections and infestations) | 2 (2)
Pneumonia (Infections and infestations) | 2 (2) — Does not Include the SAEs
Sinusitus (Infections and infestations) | 3 (3)
Upper Respiratory Infection (Infections and infestations) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 6 (6)
Contusion (Injury, poisoning and procedural complications) | 3 (3)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 4 (4)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Headache (Nervous system disorders) | 7 (7)
Hypoasthesia (Nervous system disorders) | 2 (2)
Myasthenia Gravis (Nervous system disorders) | 6 (6) — Does not include SAEs
Paraesthesia (Nervous system disorders) | 14 (14)
Depression (Nervous system disorders) | 2 (2)
Insomnia (Nervous system disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 3 (3)

LIMITATIONS AND CAVEATS:
The study was terminated due to lack of measure appropriate data. The analysis of the MG-ADL score was removed in Statistical Analysis Plan (SAP), dated 21FEB2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (5):
  • Study Protocol: Original Protocol (2017-11-12): https://cdn.clinicaltrials.gov/large-docs/66/NCT03579966/Prot_000.pdf
  • Study Protocol: Amendment 1 (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/66/NCT03579966/Prot_001.pdf
  • Statistical Analysis Plan: Version 1 PBRS (2022-10-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03579966/SAP_002.pdf
  • Statistical Analysis Plan: Version 1 StatKing (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/66/NCT03579966/SAP_003.pdf
  • Statistical Analysis Plan: version 2.0 PBRS (2023-02-21): https://cdn.clinicaltrials.gov/large-docs/66/NCT03579966/SAP_004.pdf